CLINICAL TRIAL: NCT02340988
Title: An Open-Label Study to Assess the Drug-Drug Interaction Potential of a Single 1200 mg IV Dose of Orbactiv (Oritavancin) Co-Administered With Warfarin in Healthy Subjects.
Brief Title: Drug-Drug Interaction Potential of Orbactiv (Oritavancin) Co-Administered With Warfarin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDCO-ORI-14-02
Record Dates: First submitted 2014-12-18; First posted 2015-01-19 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Healthy
MeSH Terms: interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oritavancin and Warfarin (Experimental): Oritavancin 1200 mg Single-Dose IV Oritavancin Diphosphate given simultaneously with 25mg dose of Warfarin
  Interventions: Drug: Single-Dose IV Oritavancin Diphosphate and Warfarin
- Warfarin 24 hours post dose (Experimental): 25mg dose of Warfarin given 24 hours post 1200 mg Single-Dose IV Oritavancin Diphosphate.
  Interventions: Drug: Single-Dose IV Oritavancin Diphosphate and Warfarin 24 hour post dose

INTERVENTIONS:
Drug: Single-Dose IV Oritavancin Diphosphate and Warfarin — Oritavancin will be administered as a single IV infusion simultaneously with Warfarin. The infusion will last approximately 3 hours.
  Other Names: Oritavancin Diphosphate
  Arms: Oritavancin and Warfarin
Drug: Single-Dose IV Oritavancin Diphosphate and Warfarin 24 hour post dose — Oritavancin will be administered as a single IV infusion and 24 hours post dose subjects will receive 25mg of Warfarin. The infusion will last approximately 3 hours.
  Other Names: Oritavancin Diphosphate
  Arms: Warfarin 24 hours post dose

SUMMARY:
The purpose of this study is to assess the drug interaction potential and time course of the effect of oritavancin on warfarin pharmacokinetics in an open label, single arm manner.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to provide written informed consent before initiation of any study-related procedures.
2. Subject is a healthy male or female adult between 18 and 55 years of age, inclusive.
3. Subject has a body mass index (BMI) < 45 kg/m^2.
4. Subject is in good health based on medical history and physical examination findings.
5. Female subject is surgically sterile, postmenopausal, or, if of childbearing potential, agrees to use at least 2 acceptable methods of birth control (e.g. prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, barrier methods, abstinence) or male partner sterilization alone for the duration of the study until 60 days after study drug administration.
6. Subject agrees to abstain from caffeine and theobromine containing products and the consumption of Seville oranges, grapefruit (including grapefruit juice), broccoli, brussels sprouts, charcoal grilled meat, and energy drinks from 48 hours before study drug administration and throughout the clinical phase of the study.

Exclusion Criteria:

1. Has any condition, including findings in the medical history or in pre-study assessments that constitutes a risk or a contraindication for the participation in the study or completing the study.
2. Positive breath test for alcohol and/or positive urine test for drugs of abuse at Screening.
3. Has a history or presence of alcohol/drug abuse within 2 years. Alcohol abuse is defined as regularly consuming >3 units/day (21 units per week for men), >2 units/day (14 drinks/week) for women. 1 unit of alcohol is defined as a can of 4% beer (330 mL), approximately 190 mL of 6-7% beer (malt liquor), a glass of 40% spirits (30 mL), or a glass of wine (100 mL).
4. Blood or plasma donation within past 2 months.
5. History of hypersensitivity to glycopeptide antibiotics (that have a similar chemical structure to oritavancin) or to any of the excipients of oritavancin.
6. History of hypersensitivity to warfarin or other 4-hydroxycoumarins, or to any of the excipients of warfarin.
7. Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 90 days prior to enrollment and/or unwilling to allow at least two months before participation in another drug trial following the current trial.
8. Treatment with any prescription or OTC (over the counter) drugs or herbal nutritional supplements within 2 weeks of Screening, with the exception of acetaminophen/paracetamol for minor headache. Subjects will not be allowed to receive medications for the duration of the study (except the above-mentioned acetaminophen/paracetamol). Birth control or other hormone replacement is also permitted as long as it has been taken at a stable dose for at least three months before the Screening Visit and remains stable for the duration of the study.
9. Females who are pregnant or nursing or who have a positive pregnancy test result at screening.
10. Males who are unwilling to practice abstinence or use an acceptable method of birth control during the entire study period (i.e. condom with spermicide)
11. Known protein C or protein S deficiency.
12. Inflammatory Bowel Disease or conditions which may decrease the absorption of warfarin.
13. History of bleeding tendencies (e.g. history of menorrhagia, gastrointestinal bleeding).
14. History of heparin-induced thrombocytopenia.
15. Surgery within the last 30 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure: Ratio of warfarin PK parameters - AUC and Cmax (area under the plasma concentration time curve and maximum plasma concentration) pre and post oritavancin dose and duration of effect. | Day 1-14
  Ratio of warfarin PK parameters - AUC and Cmax (area under the plasma concentration time curve and maximum plasma concentration) pre and post oritavancin dose and duration of effect.

SECONDARY OUTCOMES:
Secondary Outcome Measures: Safety of the administration of warfarin and oritavancin will be assessed according to clinical laboratory parameters, and adverse events (AEs) and serious adverse events | Day 1 through Day 21
  Safety of the administration of warfarin and oritavancin will be assessed according to clinical laboratory parameters, and adverse events (AEs) and serious adverse events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanabria, MD, Principal Investigator — Spaulding Clinical
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States